CLINICAL TRIAL: NCT05617105
Title: Molecular Characterization of Perivascular Epithelioid Cell Tumors
Acronym: PEComesCells
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7550
Record Dates: First submitted 2022-11-07; First posted 2022-11-15 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Perivascular Epithelioid Cell Tumor, Malignant
Keywords: Perivascular epithelioid cell tumors; PEComas; Myomelanocytic markers; Angiomyolipomas; Lymphangioleiomyomatoses; Visceral tumors; Fluorescence In Situ Hybridization
MeSH Terms: conditions — Perivascular Epithelioid Cell Neoplasms; Angiomyolipoma; Lymphangioleiomyomatosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Perivascular epithelioid cell tumors (PEComas) are rare and are characterized by the expression of myomelanocytic markers. They are a complex family that includes angiomyolipomas, lymphangioleiomyomatoses and other soft tissue and visceral tumors. Due to the low prevalence of these tumors, the natural history is unclear; furthermore, a molecular classification integrating clinical, pathological and molecular parameters has not been described to date.

ELIGIBILITY:
Inclusion criteria:

* Major patient (≥18 years)
* Minor patient (1 to 17 years old)
* PEComas diagnosed in France between 01/01/1990 and 15/09/2019 and reviewed by a sarcoma referral pathologist

Exclusion criteria :

* Opposition of the patient (or the holders of parental authority) to participate in the study
* Biological tissue from a patient who does not meet all the inclusion criteria
* Classic triphasic angiomyolipoma or lymphangioleiomyomatosis
* Inability to provide informed information to the subject
* Patient under court protection
* Patient under guardianship or curatorship

Min Age: 1 Year | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: patients having PEComas diagnosed in France between 01/01/1990 and 15/09/2019 and reviewed by a sarcoma referral pathologist
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
To retrospectively describe the percentage of tumors with FISH (Fluorescence In Situ Hybridization) identification of the TFE3 rearrangement out of 100 cases of PEComas diagnosed in France between 01 January 1990 and 15 September 2019 | Files analysed retrospectively from January 01, 1990 to September 15, 2019 will be examined

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'Oncologie - CHU de Strasbourg - France, Strasbourg, France